CLINICAL TRIAL: NCT06691568
Title: Effectiveness of an Air Purifier on Asthmatic and Cat-allergic Subjects in the ALYATEC Environmental Exposure Chamber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dyson Technology Ltd (Industry)
Collaborators: Alyatec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 664E-BP06-001
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Cat Allergy
Keywords: Cat allergy; EAR; Asthma; Purifier
MeSH Terms: conditions — Asthma | interventions — Air Filters

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Purifiers were active during cat allergen exposure
  Interventions: Device: Air purifier
- Placebo (Placebo Comparator): Purifiers were inactive during cat allergen exposure
  Interventions: Device: Air purifier

INTERVENTIONS:
Device: Air purifier — Purifiers were turned on for the active group and off for the placebo

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of air purifiers in reducing allergy symptoms in patients with a cat allergy. The main question it aims to answer is:

If there is a reduction of early asthmatic response (EAR) compared to placebo.

Participants were asked to remain in an exposure chamber for 2 hours while their symptoms were monitored.

DETAILED DESCRIPTION:
For this protocol, 30 patients with cat allergies were exposed to 80ng/m3 of Fel d 1 allergen in the ALYATEC Environmental Exposure Chamber (EEC).

The active group of 15 had Dyson BP06 air purifiers running at speed 2, while the placebo group had the purifiers on, but not circulating air (speed 0). Participants were monitored for the primary objective of reduction of EAR, alongside other secondary objectives:

1. To evaluate the efficacy of air purifier on time to induce EAR during a 2-hour cat allergen exposure in ALYATEC EEC compared to placebo
2. To evaluate the efficacy of air purifier on allergic rhino-conjunctivitis symptoms during a 2-hour cat allergen exposure in ALYATEC EEC compared to a placebo
3. To evaluate the efficacy of air purifier on bronchial response severity during a 2-hour cat allergen exposure in ALYATEC EEC compared to placebo.
4. To evaluate the rescue treatments used after 2-hour cat allergen exposure with the air purifier compared to placebo
5. To evaluate the efficacy of air purifier on allergic rhinitis symptoms during a 2-hour cat allergen exposure in ALYATEC EEC compared to a placebo

ELIGIBILITY:
Inclusion Criteria:

* Subjects who signed the written informed consent
* Men or women aged between 18- and 65-year-old
* Subjects covered by health social identification number
* Subjects able to understand and complete study-related procedures
* Subjects reported history of symptomatic cat allergen-triggered asthma (GINA1-2) with or without associated allergic rhinitis and/or conjunctivitis
* Positive skin prick test (SPT) with cat hair extract with mean wheal diameter ≥ 5 mm compared to negative control (NaCl reaction < 2 mm)
* Subjects with FEV1≥70% predicted at screening and before allergen exposure,
* Subjects with at least one drop in FEV1 ≥ 20% within the 2- hours exposure at baseline (V2)
* Women of childbearing potential with a negative pregnancy test throughout the study period and highly effective contraception: oral contraceptives, condom with spermicide, intrauterine device, bilateral tubal ligation, vasectomized partner.

Exclusion Criteria:

* Allergen immunotherapy to cat allergen for more than 1 month in the 3 years prior to the screening visit
* Ongoing allergen immunotherapy to another allergen
* History of anaphylactic reactions to cat allergen exposure or cat allergen immunotherapy
* History of anaphylactic reactions to another allergen in the last 6 weeks before inclusion
* Nasal polyposis, deviation of nasal septum, or diagnosis of uncontrolled non- allergic rhinitis
* Subjects allergic to indoor environmental allergens (molds, house dust mite allergens) with obvious exposure to these allergens causing allergic symptoms
* No cat exposure at home for the past year and must continue having no exposure at home during the study; cat exposure outside of the home shall be avoided for at least one week prior to any Cat Allergen Challenge
* Subjects with pollen season allergies (birch, grass, ash) will not be able to participate in the study during the pollen season for these allergens
* Conjunctival diseases such as severe keratitis, or other ocular disorders, ocular pain and/or photophobia during pollen season
* Moderate to severe asthma GINA 3 to 5

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
To measure the efficacy of air purifier on reducing the frequency of early asthmatic response (EAR) during a 2-hour cat allergen exposure in ALYATEC EEC compared to placebo. | Within the 2 hour exposure period
  Comparing the number of subjects with a drop in FEV1≥ 20% within the 2-hour exposure

SECONDARY OUTCOMES:
To evaluate the efficacy of air purifier on time to induce EAR during a 2-hour cat allergen exposure in ALYATEC EEC compared to placebo | Within the 2 hour exposure period
To evaluate the efficacy of air purifier on allergic rhino-conjunctivitis symptoms during a 2-hour cat allergen exposure in ALYATEC EEC compared to a placebo | Within the 2 hour exposure period

OTHER OUTCOMES:
To evaluate the efficacy of air purifier on bronchial response severity during a 2-hour cat allergen exposure in ALYATEC EEC compared to placebo | Within the 2 hour exposure period
To evaluate the rescue treatments used after 2-hour cat allergen exposure with the air purifier compared to placebo | Within the 2 hour exposure period
To evaluate the efficacy of air purifier on allergic rhinitis symptoms during a 2-hour cat allergen exposure in ALYATEC EEC compared to a placebo | Within the 2 hour exposure period

CONTACTS AND LOCATIONS:
Locations (1):
- ALYATEC - Nouvel Hôpital Civil, Strasbourg, France